CLINICAL TRIAL: NCT02396251
Title: A Multi-Centre, Evaluator-Blinded Study to Evaluate Efficacy and Safety of R Volumizer for Cheek Augmentation
Brief Title: Evaluation of Efficacy and Safety of Hyaluronic Acid (HA) Product for Cheek Augmentation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor business reasons
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43VZ1407
Record Dates: First submitted 2015-02-27; First posted 2015-03-24 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2019-09

CONDITIONS: Facial Tissue Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA experimental (Experimental): HA experimental only
  Interventions: Device: HA experimental
- HA comparator (Active Comparator): HA experimental + HA comparator
  Interventions: Device: HA experimental; Device: HA comparator

INTERVENTIONS:
Device: HA experimental
Device: HA comparator
  Arms: HA comparator

SUMMARY:
A multi-centre, evaluator-blinded study in subjects undergoing cheek augmentation. The study is designed to assess efficacy with regard to aesthetic midface augmentation and safety after treatment with HA product.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed and dated informed consent to participate in the study including release of copyright of images
* Man or woman aged 18 years or older
* Be willing to abstain from any other facial plastic surgical or cosmetic procedures in close proximity to the treated area

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable HA gel
* History of bleeding disorder or treatment with anticoagulants, thrombolytics, or inhibitors of platelet aggregation, omega-3, or vitamin E within 2 weeks before treatment
* Treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy, topical retinoids, systemic or topical corticosteroids within 3 months before treatment and systemic retinoids within 6 months before treatment
* Previous tissue augmenting therapy or contouring with permanent filler, fat-injection or permanent implant placed in the area to be treated
* The subject is, in the opinion of the investigator, unlikely to comply with the clinical investigational plan or is unsuitable for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (2):
- Sweden (2):
  - Gothenburg
  - Stockholm

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Both Cheeks Group: HA product under investigation in both cheeks
- Split-face Group: HA product under investigation in one cheek and a comparator in the other cheek.
Period: Overall Study
Arm/Group | Both Cheeks Group | Split-face Group
Started | 36 | 12
Completed | 23 | 7
Not Completed | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Both Cheeks Group | Split-face Group | Total
Number analyzed (Participants) | 36 | 12 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 11 | 46
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11) | 44.8 (10.2) | 42 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 12 | 46
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 35 | 11 | 46
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 36 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders in Midface Fullness Using Photo Scale
Description: Evaluation of midface fullness, determined by the percentage of responders at 3 months after last treatment, in both cheeks, derived from the Blinded Evaluator's live assessment of a validated photo scale. A responder was defined as a subject with ≥1 grade improvement from baseline in both cheeks.
Time Frame: 3 months
Population: The primary objective applied to the group treated with the investigational HA product in both cheeks.
  Only exploratory objective applied to the split-face group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Both Cheeks Group: Subjects with at least 1 step improvement on validated photo scale in both cheeks as assessed by the Blinded evaluator, Both cheeks group
Arm/Group | Both Cheeks Group
Number analyzed (Participants) | 31
percentage of participants | 93.5 [78.6 to 99.2]

2. Secondary Outcome: Percentage of Responders in Midface Fullness Using Photo Scale
Description: Evaluate midface fullness as determined by percentage of responders at 4 weeks and 6, 9, 12 and, if applicable, 15 months after last treatment as well as 4 weeks and 3 months after re-treatment, derived from the Blinded Evaluator's live assessment of photo scale. A responder was defined as a subject with ≥1 grade improvement from baseline in both cheeks.
Time Frame: 15 months
Population: Number of participants with available data varied during the study. The secondary objective applied to the group treated with the investigational HA product in both cheeks.
  Only exploratory objective applied to the split-face group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Both Cheeks Group
Number analyzed (Participants) | 34
percentage of participants
  4 weeks after last treatment | 88.2 [72.5 to 96.7]
  3 months: number analyzed (Participants) | 31
  3 months | 93.5 [78.6 to 99.2]
  6 months: number analyzed (Participants) | 30
  6 months | 90 [73.5 to 97.9]
  9 months: number analyzed (Participants) | 27
  9 months | 81.5 [61.9 to 93.7]
  12 months: number analyzed (Participants) | 30
  12 months | 43.3 [25.5 to 62.6]
  15 months: number analyzed (Participants) | 20
  15 months | 25 [8.7 to 49.1]
  4 weeks after re-treatment: number analyzed (Participants) | 5
  4 weeks after re-treatment | 100 [47.8 to 100]
  3 months after re-treatment: number analyzed (Participants) | 4
  3 months after re-treatment | 100 [39.8 to 100]

ADVERSE EVENTS:
Time Frame: 2 years, 9 months (from first subject screening to last subject's last visit).
Description: Groups for each intervention separately cannot be provided since most of the Adverse Events (AEs) are not related to study product. Analysis groups were "Both cheeks group" and "Split-face group" (as presented here). In the Split-face group, only two AEs were assessed as related to study product/device injection procedure: the AE "Implant site pain" which was assessed as related to the HA product under investigation, and the AE "Eye pain" which was not assessed as related to a specific product.
Arm/Group | Both Cheeks Group | Split-face Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/36 | 1/12
Other Adverse Events (participants affected / at risk) | 23/36 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Both Cheeks Group (N=36) | Split-face Group (N=12)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Elevated TNT (Investigations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Unstable patella (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Scar left cheek (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Both Cheeks Group (N=36) | Split-face Group (N=12)
Injection site oedema (General disorders) | 2 (3) | 0 (0)
Injection site pain (General disorders) | 5 (8) | 0 (0)
Injection site swelling (General disorders) | 7 (21) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Implant site swelling (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dark circles under eyes (Eye disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes